CLINICAL TRIAL: NCT06517719
Title: Real-world Experience With Lutetium (177Lu) Vipivotide Tetraxetan in Metastatic Castration Resistant Prostate Cancer, an Observational, Multicenter, Prospective Cohort Study
Brief Title: Real-world Experience With Lutetium Vipivotide Tetraxetan in Metastatic Castration Resistant Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAAA617A1DE04
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
Keywords: metastatic castration resistant prostate cancer; mCRPC; Prostate cancer; lutetium vipivotide tetraxetan; 177Lu
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lutetium; Lutetium-177

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Lutetium (177Lu) vipivotide tetraxetan: Patients with mCRPC initiating lutetium (177Lu) vipivotide tetraxetan
  Interventions: Other: lutetium (177Lu) vipivotide tetraxetan

INTERVENTIONS:
Other: lutetium (177Lu) vipivotide tetraxetan — This is an observational study. There is no treatment allocation. The decision to initiate lutetium vipivotide tetraxetan will be based solely on clinical judgement.

SUMMARY:
The purpose of this study is to describe routine clinical practice with lutetium (177Lu) vipivotide tetraxetan on Health related quality of life (HRQoL) at baseline, on treatment, and post progression.

DETAILED DESCRIPTION:
This non-interventional observational, prospective cohort study is using primary data collection to describe the routine clinical practice and HRQoL of patients with Metastatic castration-resistant prostate cancer (mCRPC) initiating lutetium (177Lu) vipivotide tetraxetan using patient questionnaires.

Data will be collected at the following time points: pre-index (if patient is eligible), index date (first application of lutetium (177Lu) vipivotide tetraxetan), during treatment, at EoT, and during follow-up.

The duration of a treatment cycle is 6 weeks (± 1 week). Patients will be treated for up to 6 cycles (as per local label).

EoT visit / assessments will be performed after the last lutetium (177Lu) vipivotide tetraxetan application.

Follow-up period: patient data will be collected if available up to 1 year after EoT.

ELIGIBILITY:
Inclusion Criteria:

All patients must meet the following inclusion criteria during the identification period:

* Adult male patients diagnosed with mCRPC and initiating lutetium (177Lu) vipivotide tetraxetan by treating physician as per local label. After treatment decision enrollment is allowed before date of cycle 1 or within 2 weeks after the date of Cycle 1.
* ≥ 18 years old at the time of enrollment
* Written informed consent must be obtained prior to any data collection
* Willing to participate in Quality of Life post treatment date collection for 1 year

Exclusion Criteria:

Patients must not meet the following exclusion criterion during the identification period:

- Simultaneous participation in any investigational trial or simultaneous participation in another Novartis-sponsored non-interventional study with lutetium (177Lu) vipivotide tetraxetan

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult male patients with mCRPC
Study Population: Adult male patients with mCRPC
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy - Prostate (FACT-P) | Baseline, up to 1 year after end of treatment
  FACT-P assesses symptoms/problems related to prostate carcinoma and its treatment. It is a combination of the FACT- General + the Prostate Cancer Subscale (PCS). The FACTGeneral (FACT-G) is a 27 item Quality of Life (QoL) measure that provides a total score as well as subscale scores: Physical (0-28), Functional (0-28), Social (0-28), and Emotional Well-being (0-24). The total score range is between 1-108, higher scores indicates better for total score and subscale scores. PCS is a 12-item prostate cancer subscale that asks about symptoms and problems specific to prostate cancer (Range 0-48, higher scores better). The FACT-P total score is the sum of all 5 subscale scores of the FACT-P questionnaire and ranges from 0-156. Higher scores indicate higher degree of functioning and better quality of life.
Change from baseline in FACT-P | Baseline, up to 1 year after end of treatment
  FACT-P assesses symptoms/problems related to prostate carcinoma and its treatment. It is a combination of the FACT- General + the Prostate Cancer Subscale (PCS). The FACTGeneral (FACT-G) is a 27 item Quality of Life (QoL) measure that provides a total score as well as subscale scores: Physical (0-28), Functional (0-28), Social (0-28), and Emotional Well-being (0-24). The total score range is between 1-108, higher scores indicates better for total score and subscale scores. PCS is a 12-item prostate cancer subscale that asks about symptoms and problems specific to prostate cancer (Range 0-48, higher scores better). The FACT-P total score is the sum of all 5 subscale scores of the FACT-P questionnaire and ranges from 0-156. Higher scores indicate higher degree of functioning and better quality of life.
Functional Assessment of Cancer Therapy-Radionuclid Therapy (FACT-RNT) | Baseline, up to 1 year after end of treatment
  The FACT-RNT (Functional Assessment of Cancer Therapy - Radionuclide Therapy) is a Patient Reported Outcomes (PRO) new measure developed using FACIT specific questions (items), selected from FACIT item bank, to assess treatment-related symptoms of special interest associated with radioligand therapies.
  The FACT-RNT contains items assessing dry mouth, dry eyes, vomiting, diarrhea, constipation, loss of appetite, fatigue, impact of fatigue, bone pain, and isolation due to illness or treatment. FACT-RNT score range 0 to 60, with higher score indicating better quality of life.
Change from baseline in FACT-RNT | Baseline, up to 1 year after end of treatment
  The FACT-RNT (Functional Assessment of Cancer Therapy - Radionuclide Therapy) is a Patient Reported Outcomes (PRO) new measure developed using FACIT specific questions (items), selected from FACIT item bank, to assess treatment-related symptoms of special interest associated with radioligand therapies.
  The FACT-RNT contains items assessing dry mouth, dry eyes, vomiting, diarrhea, constipation, loss of appetite, fatigue, impact of fatigue, bone pain, and isolation due to illness or treatment. FACT-RNT score range 0 to 60, with higher score indicating better quality of life.
Brief Pain Inventory-Short Form (BPI-SF) | Baseline, up to 1 year after end of treatment
  The BPI-SF is a publicly available instrument to assess the pain and includes severity and interference scores. BPI-SF is an 11-item selfreport questionnaire that is designed to assess the severity and impact of pain on daily functions of a participant. Pain severity score is a mean value for BPI-SF questions 3, 4, 5 and 6 (questions inquiring about the extent of pain, where the extent is ranked from 0 [no pain] to 10 [pain as bad as you can imagine]). Pain severity progression is defined as an increase in score of 30% or greater from baseline without decrease in analgesic use
Change from baseline in BPI-SF | Baseline, up to 1 year after end of treatment
  The BPI-SF is a publicly available instrument to assess the pain and includes severity and interference scores. BPI-SF is an 11-item selfreport questionnaire that is designed to assess the severity and impact of pain on daily functions of a participant. Pain severity score is a mean value for BPI-SF questions 3, 4, 5 and 6 (questions inquiring about the extent of pain, where the extent is ranked from 0 [no pain] to 10 [pain as bad as you can imagine]). Pain severity progression is defined as an increase in score of 30% or greater from baseline without decrease in analgesic use
Radiographic progression | Up to 1 year after end of treatment
  Radiographic progression is measured with radiographic imaging (e.g. CT with contrast/MRI, bone scan, PET/CT, SPECT/CT) according to RECIST/PCWG3
Clinical progression | Up to 1 year after end of treatment
  Unequivocal clinical progression (UCP) is considered a worsening of clinical status with or without radiographic progression (RAD): escalation in cancer related-pain, immediate need for initiation of new anticancer treatment, surgical, or radiological intervention, deterioration in ECOG to grade 3 or higher, in the opinion of investigator
Time to prostate-specific antigen (PSA) progression | Up to 1 year after end of treatment
  Time to PSA progression is defined as time from randomization to first PSA progression.
  PSA progression is defined as the date that a ≥ 25% increase in PSA and an absolute increase of 2 ng/mL or more from the nadir or baseline is documented and confirmed by a second consecutive value obtained 3 or more weeks later. Rises in PSA within the first 12 weeks will be ignored in the absence of other evidence of disease progression (adapted from Prostate Cancer Working Group (PCWG3) Guidance).
Prostate-specific antigen (PSA) 30/50/90 | Up to 1 year after end of treatment
  Response rates are defined as the proportion of patients who have a ≥30%/50%/90% decrease in PSA from baseline that is confirmed by a second PSA measurement.
Progression-free survival (PFS) | Up to 1 year after end of treatment
  PFS, defined as the time from initial treatment to the first documented disease progression or death due to any cause, whichever occurs first.
Progression-free survival 2 (PFS2) | Up to 1 year after end of treatment
  PFS2, defined as time from initial treatment to the first documented disease progression or death under the treatment after lutetium (177Lu) vipivotide tetraxetan.
Overall Survival (OS) | Up to 1 year after end of treatment
  OS defined as the time from initial treatment until death from any cause.
Time to initiation of pain medication | Up to 1 year after end of treatment
  Time to initiation of pain medication is defined as time from index date to the first use of any pain medication or progression.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (32):
- Germany (32):
  - Novartis Investigative Site, Konstanz, Baden-Wurttemberg
  - Novartis Investigative Site, Stuttgart, Baden-Wurttemberg
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Cottbus, Brandenburg
  - Novartis Investigative Site, Frankfurt (Oder), Brandenburg
  - Novartis Investigative Site, Ludwigshafen, Germany
  - Novartis Investigative Site, Marburg, Hesse
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Fulda
  - Novartis Investigative Site, Herford
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Trier
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm

IPD SHARING:
Plan to Share IPD: No